CLINICAL TRIAL: NCT00692224
Title: Effect of Oral Zinc Given Daily Between Days 2 and 7 of Life to Term or Near Term Neonates With Serum Bilirubin Levels of More Than 6 mg/dL at 24 ± 6 Hours of Life on Hyperbilirubinemia and Phototherapy
Brief Title: Efficacy of Zinc in Reducing Hyperbilirubinemia Among High Risk Neonates - A Double Blind Randomized Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Nidhi Rana, All India Institute of medical sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A-68:12/08/2005
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Neonatal Jaundice
Keywords: neonatal jaundice; zinc; hyperbilirubinemia; enterohepatic circulation; bilirubin
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): study group received zinc gluconate in a dose of 10 mg/day
  Interventions: Drug: zinc gluconate
- 2 (Placebo Comparator): placebo group received placebo which was identical in color, taste and appearance and packaged in similar looking bottles.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zinc gluconate — zinc gluconate syrup - 10mg/day in two divided doses from day 2 to day 7 of life
  Arms: 1
Drug: placebo — placebo was packed in similar looking bottles and ad similar taste as zinc gluconate drug
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of 10 mg of oral zinc given daily between days 2 and 7 of life to term or near term neonates with serum bilirubin levels of more than 6 mg/dL at 24 ± 6 hours of life on hyperbilirubinemia and phototherapy.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia is a common problem occurring in nearly 5-25% neonates.Inhibition of enterohepatic circulation is one of the therapies being tried for neonatal jaundice. Studies have suggested that in a neonate, the postulated enterohepatic pathway is of a magnitude that could be significant in the overall body economy of bilirubin.Zinc has also been investigated for its role in decreasing the STB levels by inhibiting enterohepatic circulation. There have been animal studies which have investigated the role of zinc in decreasing the serum bilirubin levels. The mechanism proposed is that zinc salts precipitate Unconjugated bilirubin from unsaturated micellar solution of bile salts and consequently inhibit the enterohepatic circulation of bilirubin. This is the first study to evaluate the role of zinc in neonatal jaundice.

Study Design: In this randomized placebo controlled clinical trial neonates born at ≥35 wk of gestation and with total serum bilirubin ≥6mg% were given either zinc gluconate (n = 148) or placebo (n = 146) in a dose of 10mg per day between days 2 and 7 of life. Jaundice was assessed clinically and total serum bilirubin estimated using spectrophotometry. Infants were followed up clinically until discharge and then again at day 7 of life. Hyperbilirubinemia was defined as total serum bilirubin ≥15mg%.

Results: Incidence of hyperbilirubinemia was comparable in zinc and placebo groups (OR 0.95, 95% CI 0.50-1.67, p=0.92). The requirement of phototherapy was similar in the two groups (OR 0.81, 95% CI 0.41-1.61, p=0.55). The mean hours of phototherapy in the zinc group were also similar in the two groups (p=0.63). No significant difference with respect to mean levels of bilirubin (mg/dL) at 72±12 hours of age was observed in two groups(zinc 11.3±3.3,placebo 11.5±3.8,p=0.63). No significant adverse effects of zinc were noted.

Conclusion: Twice daily zinc administration in a dose of 10 mg/day does not reduce hyperbilirubinemia in at risk neonates in the first week of life.

.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born at ≥35 weeks gestation and with total serum bilirubin ≥ 6 mg/dL at 24±6 h of life.

Exclusion Criteria:

* Rh incompatibility
* Those given exchange transfusion/ phototherapy within 24 h of age.
* Major gross congenital anomaly
* Anticipated to require neonatal intensive care or required neonatal intensive care for more than 24 h.
* Systemic sepsis

Ages: 18 Hours to 30 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 294 (Actual)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperbilirubinemia defined as total serum bilirubin more than or equal to 15 mg/dL at anytime between days 2 and 7 of life. | first week of life

SECONDARY OUTCOMES:
The mean total serum bilirubin level at 72±12 hours of age. | first two weeks of life
The proportion of infants requiring phototherapy and the duration thereof | first two weeks of life

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Rana, M.D, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute Of Medical Sciences, New Delhi, National Capital Territory of Delhi, India